CLINICAL TRIAL: NCT04877470
Title: Baseline-characteristics of Patients Referred to a Secondary Spine Centre
Acronym: CHAPARS
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: Z2021026
Record Dates: First submitted 2021-04-22; First posted 2021-05-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Spine Disease; Characteristics Disease; Spinal Disease; Demography
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly referred patients visiting the spine-centre: Newly referred patients visiting the spine-centre at Zuyderland Medical Centre Heerlen in 2019, from 01.01.2019 until 31.12.2019.
  Interventions: Other: Consultation at spine-centre

INTERVENTIONS:
Other: Consultation at spine-centre — All patients who visited the spine-centre for the first time in 2019 are included in this group.

SUMMARY:
A retrospective cohort study will be conducted in Zuyderland Medical Centre Heerlen, the Netherlands. All patients that were referred to the spine-centre between 01.01.2019 and 31.12.2019 will be included for analysis.

This study aims to evaluate baseline characteristics, including baseline questionnaires, and information about the given treatments for all patients referred to the spine centre.

DETAILED DESCRIPTION:
The incidence of back and neck pain is increasing in our ageing population. Back pain is amongst the conditions with the highest burden of disease in terms of years lived with disability (YLD). The majority of people experiences at least one period of back pain in their lifetime. The incidence of back complaints increases with age. Due to ageing of the population, the number of patients with back pain exponentially increases. Since 1980, the global population of people older than 60 years has doubled and this number is expected to double again by 2050. Patients with back or neck pain and/or symptoms of radiculopathy, and suspected spinal pathology, are often referred to a secondary spine centre. A large number of these patients will receive conservative treatment and only a small number eventually receives a surgical intervention. There is a broad array of conservative treatment options, including medication, manipulative care, physical therapy, treatment by pain specialists, and rehabilitation. The increasing incidence of spinal pathologies likewise leads to an increase in spinal surgeries. The ageing population is one of the most prominent factors by which the number of spine surgeries has increased and will even increase further in the future. Previous studies concerning the national US bill for spine related care in 2006 estimated that direct medical expenditures were over $85 billion. Over the last decades, the costs of spine related healthcare have increased at an alarming rate and will even increase further. To limit the increase of healthcare-related costs concerning spine-related healthcare in an ageing population, the selection and profiling of subgroups of patients requiring different types of treatment should be ameliorated to optimize spinal care. To date, adequate knowledge on baseline characteristics is lacking, and thereby insufficient to perform patient profiling.

This study aims to evaluate baseline characteristics, including baseline questionnaires, and information about the given treatments for all patients referred to the spine centre. Insight in the specific characteristics of different patient groups, for example different types of conservative interventions or conservative versus surgical interventions, could provide a valuable insight during counselling.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred patients visiting the spine-centre at Zuyderland Medical Centre Heerlen in 2019, from 01.01.2019 until 31.12.2019.
* Minimum age of 18 years.
* Documented treatment (surgical or conservative).

Exclusion Criteria:

* Documented objection to participate in scientific research.
* No baseline questionnaires available

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients who are referred to the spine-centre at Zuyderland Medical Centre
Sampling Method: Probability Sample
Enrollment: 4855 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Age | 01.01.2019-31.12.2019
  Age in years.
Gender | 01.01.2019-31.12.2019
  Male, female, other
Body Mass Index (BMI) | 01.01.2019-31.12.2019
  BMI = kg/m2
Smoking (current status) | 01.01.2019-31.12.2019
  Yes/no
Duration of symptoms | 01.01.2019-31.12.2019
  Time since onset of symptoms in months.
Type of complaints | 01.01.2019-31.12.2019
  Back pain, leg pain, arm pain or neck pain
Diagnosis | 01.01.2019-31.12.2019
  Final diagnosis as mention in the patient file, e.g. lytic spondylolisthesis, herniated disc etc.
History of spinal surgery | 01.01.2019-31.12.2019
  Spinal surgeries in the past, as mentioned in the patient file, e.g. lumbar interbody fusion, discectomy, etc.
Use of pain medication | 01.01.2019-31.12.2019
  Paracetamol, NSAID, opioid, neuropathic pain medication
Reason for referral | 01.01.2019-31.12.2019
  Reason for referral, as mentioned in the general practitioner's file, e.g. persistent back pain, leg pain, etc.
Diagnostics tests carried out | 01.01.2019-31.12.2019
  Diagnostics as mentioned in the patient file, e.g. MRI, CT-scan, X-ray, EMG, etc.
Number of consultations | 01.01.2019-31.12.2019
  Number of consultations at the spine-centre since referral.
Follow-up period | 01.01.2019-31.12.2019
  Time between the first consultation and the last follow-up consultations, in months.

SECONDARY OUTCOMES:
EuroQol 5D | 01.01.2019-31.12.2019
  Score per item, total score is based on Value Sets. A lower score indicated a better quality of life.
Roland Disability Questionnaire | 01.01.2019-31.12.2019
  Score: 0-24. A higher score indicated more disability.
Tampa Scale of Kinesiophobia | 01.01.2019-31.12.2019
  Score: 17-68. 17 means no kinesiophobia, 68 means severe kinesiophobia
Visual Analogue Scale (VAS) | 01.01.2019-31.12.2019
  Score: 0-10. 0 is no pain, 10 is maximum pain
Western Ontario and McMaster Universities Osteoarthritis Index | 01.01.2019-31.12.2019
  Score: 0-96. A higher score indicates more complaints and disability.
Oxford Hip Score | 01.01.2019-31.12.2019
  Score: 12-60. Item scores are summed to give a total score from anywhere between 12 and 60. The lower the score, the better the outcome.
Oswestry Disability Index | 01.01.2019-31.12.2019
  Score: 0-100 . A higher scores indicated more disability.
Örebro Musculoskeletal Pain Screening Questionnaire | 01.01.2019-31.12.2019
  Score: 0-210. A higher score indicated more complaints and more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Anouk Smeets, MD, PhD, Principal Investigator — Zuyderland Medisch Centrum
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Deis N, Findlay JM. Appropriateness of lumbar spine referrals to a neurosurgical service. Can J Neurol Sci. 2010 Nov;37(6):843-8. doi: 10.1017/s0317167100051544. PMID 21059549
- [Background] Deyo RA, Mirza SK, Turner JA, Martin BI. Overtreating chronic back pain: time to back off? J Am Board Fam Med. 2009 Jan-Feb;22(1):62-8. doi: 10.3122/jabfm.2009.01.080102. PMID 19124635
- [Background] Saifi C, Cazzulino A, Laratta J, Save AV, Shillingford JN, Louie PK, Pugely AJ, Arlet V. Utilization and Economic Impact of Posterolateral Fusion and Posterior/Transforaminal Lumbar Interbody Fusion Surgeries in the United States. Global Spine J. 2019 Apr;9(2):185-190. doi: 10.1177/2192568218790557. Epub 2018 Aug 15. PMID 30984499
- [Background] de Kunder SL, Rijkers K, Caelers IJMH, de Bie RA, Koehler PJ, van Santbrink H. Lumbar Interbody Fusion: A Historical Overview and a Future Perspective. Spine (Phila Pa 1976). 2018 Aug;43(16):1161-1168. doi: 10.1097/BRS.0000000000002534. PMID 29280929
- [Background] Martin BI, Deyo RA, Mirza SK, Turner JA, Comstock BA, Hollingworth W, Sullivan SD. Expenditures and health status among adults with back and neck problems. JAMA. 2008 Feb 13;299(6):656-64. doi: 10.1001/jama.299.6.656. PMID 18270354
- [Background] Weiner DK, Kim YS, Bonino P, Wang T. Low back pain in older adults: are we utilizing healthcare resources wisely? Pain Med. 2006 Mar-Apr;7(2):143-50. doi: 10.1111/j.1526-4637.2006.00112.x. PMID 16634727